CLINICAL TRIAL: NCT04053959
Title: A Study to Assess the Effect and Safety of Artificial Intelligence Assisted Insulin Titration System on Glucose Control in Type 2 Diabetes Mellitus Patients: A Single-center, Open-labeled, Parallel, Randomized Controlled Trial
Brief Title: Artificial Intelligence Assisted Insulin Titration System
Acronym: iNCDSS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZSE-201902
Record Dates: First submitted 2019-08-10; First posted 2019-08-13 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: A paralle group, randomized, controlled study to assess the effect and safety of artificial intelligence assisted insulin dosage titration system on glucose control in type 2 diabetic patients
Who Masked: Participant, Outcomes Assessor
Masking Description: The research assistants who collect study outcome data will be masked to participants' intervention assignment. In addition, the adjudicators for end-points will not be aware of study-group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI Group (Experimental): Artificial intelligence assisted insulin titration system group
  Interventions: Drug: AI assisted insulin system
- Control Group (Active Comparator): Physicians decided insulin titration group
  Interventions: Drug: Physician based insulin regime

INTERVENTIONS:
Drug: AI assisted insulin system — The patients receive the insulin regime set by AI assisted insulin titration system
  Arms: AI Group
Drug: Physician based insulin regime — Patients receive the insulin regime recommended by physicians
  Arms: Control Group

SUMMARY:
This is a single-center, open-labeled, parallel group, randomized controlled trial to access the effect and safety of the Artificial Intelligence Assisted Insulin Titration System in patients with Type 2 Diabetes Mellitus.

DETAILED DESCRIPTION:
The study enrolls 44 patients with Type 2 Diabetes in Zhongshan Hospital who are on treatment with insulin for at least 3 months. They are randomly allocated into 2 groups at a ratio of 1:1 after screening for the inclusion and exclusion criteria. Patients in the Intervention group receive insulin regimen set by the AI assisted system and patients in Control group receive insulin regimen set by physicians. This study will be conducted in the Department of Endocrinology, Zhongshan Hospital,Fudan University and consist of a 7-day intervention period. Patient allocation will be stratified by HbA1c, BMI and previous total insulin doses.The primary endpoint is the percentage of time of sensor glucose measurements in targeted range (3.9-10 mmol/L) during the 7-days trial period.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18-75 years old;
* Subjects who had been diagnosed with type 2 diabetes;
* Subjects who are on treatment with insulin for at least 3 months;
* HbA1c: 7.0%-11.0%.

Exclusion Criteria:

* Subjects with acute complications of diabetes such as ketoacidosis or hyperglycemic hyperosmolar state;
* Subjects who change the insulin regimens during hospitalization;
* BMI ≥ 45kg/m2;
* Women who are pregnant or nursing;
* Subjects with severe cardiac, hepatic, renal or general diseases;
* Subjects with psychiatric disorders or impaired cognitive function;
* Subjects with severe edema, infections or peripheral circulation disorders;
* Patients treated with surgery during hospitalization;
* Subjects that are, in the judgement of the investigator, unlikely to comply with the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-09-27 (Actual); Primary Completion 2020-01-22 (Actual); Study Completion 2020-04-15 (Actual)

PRIMARY OUTCOMES:
Proportion of time in target range | During 7-day intervention
  The well-controlled blood glucose level is defined as the time of sensor glucose measurements in targeted range (3.9-10 mmol/L)

SECONDARY OUTCOMES:
Proportion of time in which the blood glucose level is over 10 mmol/L | During 7-day intervention
  The poor control of blood glucose level is defined as greater than 10 mmol/L
Proportion of time in which the blood glucose level is below 3.9 mmol/L | During 7-day intervention
  The hypoglycemia is defined as blood glucose level less than 3.9mmol/L
Total insulin dose | Each day during 7-day intervention
  The total insulin dose is defined as daily insulin dose

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoying Li, MD, Principal Investigator — Fudan University
Locations (1):
- 180 Fenglin Road, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xu Y, Wang L, He J, Bi Y, Li M, Wang T, Wang L, Jiang Y, Dai M, Lu J, Xu M, Li Y, Hu N, Li J, Mi S, Chen CS, Li G, Mu Y, Zhao J, Kong L, Chen J, Lai S, Wang W, Zhao W, Ning G; 2010 China Noncommunicable Disease Surveillance Group. Prevalence and control of diabetes in Chinese adults. JAMA. 2013 Sep 4;310(9):948-59. doi: 10.1001/jama.2013.168118. PMID 24002281
- [Background] Wang T, Xu Y, Xu M, Wang W, Bi Y, Lu J, Dai M, Zhang D, Ding L, Xu B, Sun J, Zhao W, Jiang Y, Wang L, Li Y, Zhang M, Lai S, Wang L, Ning G. Awareness, treatment and control of cardiometabolic disorders in Chinese adults with diabetes: a national representative population study. Cardiovasc Diabetol. 2015 Feb 26;14:28. doi: 10.1186/s12933-015-0191-6. PMID 25848699
- [Background] Ji LN, Lu JM, Guo XH, Yang WY, Weng JP, Jia WP, Zou DJ, Zhou ZG, Yu DM, Liu J, Shan ZY, Yang YZ, Hu RM, Zhu DL, Yang LY, Chen L, Zhao ZG, Li QF, Tian HM, Ji QH, Liu J, Ge JP, Shi LX, Xu YC. Glycemic control among patients in China with type 2 diabetes mellitus receiving oral drugs or injectables. BMC Public Health. 2013 Jun 21;13:602. doi: 10.1186/1471-2458-13-602. PMID 23800082
- [Background] Davies M, Storms F, Shutler S, Bianchi-Biscay M, Gomis R; ATLANTUS Study Group. Improvement of glycemic control in subjects with poorly controlled type 2 diabetes: comparison of two treatment algorithms using insulin glargine. Diabetes Care. 2005 Jun;28(6):1282-8. doi: 10.2337/diacare.28.6.1282. PMID 15920040
- [Background] Oyer DS, Shepherd MD, Coulter FC, Bhargava A, Brett J, Chu PL, Trippe BS; INITIATEplus Study Group. A(1c) control in a primary care setting: self-titrating an insulin analog pre-mix (INITIATEplus trial). Am J Med. 2009 Nov;122(11):1043-9. doi: 10.1016/j.amjmed.2008.12.026. PMID 19854333
- [Background] Yang W, Zhu L, Meng B, Liu Y, Wang W, Ye S, Sun L, Miao H, Guo L, Wang Z, Lv X, Li Q, Ji Q, Zhao W, Yang G. Subject-driven titration of biphasic insulin aspart 30 twice daily is non-inferior to investigator-driven titration in Chinese patients with type 2 diabetes inadequately controlled with premixed human insulin: A randomized, open-label, parallel-group, multicenter trial. J Diabetes Investig. 2016 Jan;7(1):85-93. doi: 10.1111/jdi.12364. Epub 2015 May 25. PMID 26816605
- [Background] Harris S, Yale JF, Dempsey E, Gerstein H. Can family physicians help patients initiate basal insulin therapy successfully?: randomized trial of patient-titrated insulin glargine compared with standard oral therapy: lessons for family practice from the Canadian INSIGHT trial. Can Fam Physician. 2008 Apr;54(4):550-8. PMID 18411384
- [Background] Rigla M, Garcia-Saez G, Pons B, Hernando ME. Artificial Intelligence Methodologies and Their Application to Diabetes. J Diabetes Sci Technol. 2018 Mar;12(2):303-310. doi: 10.1177/1932296817710475. Epub 2017 May 25. PMID 28539087
- [Background] Ashrafzadeh S, Hamdy O. Patient-Driven Diabetes Care of the Future in the Technology Era. Cell Metab. 2019 Mar 5;29(3):564-575. doi: 10.1016/j.cmet.2018.09.005. Epub 2018 Sep 27. PMID 30269984
- [Background] Thabit H, Hartnell S, Allen JM, Lake A, Wilinska ME, Ruan Y, Evans ML, Coll AP, Hovorka R. Closed-loop insulin delivery in inpatients with type 2 diabetes: a randomised, parallel-group trial. Lancet Diabetes Endocrinol. 2017 Feb;5(2):117-124. doi: 10.1016/S2213-8587(16)30280-7. Epub 2016 Nov 9. PMID 27836235
- [Background] Bally L, Thabit H, Hartnell S, Andereggen E, Ruan Y, Wilinska ME, Evans ML, Wertli MM, Coll AP, Stettler C, Hovorka R. Closed-Loop Insulin Delivery for Glycemic Control in Noncritical Care. N Engl J Med. 2018 Aug 9;379(6):547-556. doi: 10.1056/NEJMoa1805233. Epub 2018 Jun 25. PMID 29940126